CLINICAL TRIAL: NCT04025697
Title: Complete Denture Tooth Movement in Digital Light Processing Versus Conventional Fabrication Techniques: A Randomized Controlled Trial
Brief Title: Complete Denture Tooth Movement in Digital Light Processing Versus Conventional Fabrication Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaymaa Belety, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Rapid Prototyping Dentures
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Rapid Prototyping in Dentures
MeSH Terms: interventions — Denture, Complete

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional CD (Placebo Comparator): A conventional Complete denture will be constructed and the amount of denture tooth movement will be measured
  Interventions: Other: Complete Denture
- Rapid Prototyped Denture (Active Comparator): A digital light processed denture will be constructed and the amount of tooth movement will be measured
  Interventions: Other: Rapid prototyped denture

INTERVENTIONS:
Other: Complete Denture — A conventional CD will be constructed
  Arms: Conventional CD
Other: Rapid prototyped denture — A 3d printed complete denture will be constructed
  Arms: Rapid Prototyped Denture

SUMMARY:
The purposes of this study are to compare the denture tooth movement, the amount of occlusal adjustment needed and the chairside time required for CAD-CAM and conventional dentures.

PICOT Format:

P: completely edentulous patients. I: Complete denture fabricated by digital light processing method. C: Complete denture fabricated by the conventional method.

O:

Primary Outcome: Denture tooth movement

Secondary outcomes:

* Amount of occlusal adjustments needed
* Chairside time T: Three months with a wash-up period of 2 weeks

ELIGIBILITY:
Inclusion Criteria:

* Age ranging from 40-70 years.
* Cooperative patients with no history of psychological diseases.
* Completely edentulous patients with types I, II and III mandibles according to McGarry et al.

Exclusion Criteria:

* Pathological changes of residual ridges
* Patients with xerostomia.
* Patients with flabby ridges.
* Temporomandibular disorders and neuromuscular disorders e.g. Parkinson's disease

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
The amount of tooth movement | 8 months
  The amount of tooth movement will be measured immediately after denture construction using the Geomagic surface matching software (Geomagic Control 2014; 3D Systems Inc.) Laser scan images of the denture obtained both after trial setup of teeth and of the final denture after being hydrated for 24 hours. Those images will be transferred into STL files that will then be superimposed using the global registration function of the software by finding 10,000 points in common between both pre and pot processing STL files.
  Measurements will be made at different points using the software and colour surface maps will be created using the 3D comparison function to display the amount and direction of tooth movement

CONTACTS AND LOCATIONS:
Overall Officials: Iman A Radi, Study Director — Cairo University